CLINICAL TRIAL: NCT05569681
Title: Comparison of Two Different Regimens of Bemiparin as a Thromboprophylaxis After Surgery in Morbidly Obese Patients: A Randomized, Outcome-assessor Blinded Trial.
Brief Title: Two Different Regimens of Bemiparin as a Thromboprophylaxis in Morbidly Obese Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, SHAHLA KAREEM ALALAF, Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMU4
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Morbid Obesity
Keywords: LMWH; Thromboprophylaxis; Non-orthopedic surgeries; Gynecological surgeries; General surgeries; Bariatric surgeries
MeSH Terms: conditions — Obesity, Morbid | interventions — bemiparin

STUDY DESIGN:
Intervention Model Description: Postsurgical morbidly obese patients will be randomized to receive 2 different doses of Bemiparin
Masking Description: outcome-assessor blinded study. Due to inherent color differences between the two types of LMWH, the treatment administration could not be fully masked. However, treatment allocation was masked from the outcome assessor from the start by using coded envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bemiparin 3500 IU (Active Comparator): Bemiparin sodium 3,500 IU anti Xa/0.2 ml solution for injection in the pre-filled syringe will be provided for each patient in one group; subcutaneously 6 hours after the surgery(orthopedic and non-orthopedic) and then daily for up to 10 days for moderate and high - risk group and for 30 days in very high risk-group patients according to Caprinin risk classification for venous thromboembolism.
  Other Name: Hibor; Laboratories Rovi Pharmaceuticals
  Interventions: Drug: Bemiparin 3500
- Bemiparin 5000 IU (Active Comparator): Bemiparin sodium 5000 IU anti Xa/0.2 ml solution for injection in the pre-filled syringe will be provided for each patient in one group; subcutaneously 6 hours after the surgery(orthopedic and non-orthopedic) and then daily for up to 10 days for moderate and high - risk group patients and 30 days in very high-risk group surgical patients according to Caprinin risk classification for venous thromboembolism.
  Other Name: Hibor; Laboratories Rovi Pharmaceuticals
  Interventions: Drug: Bemiparin 5000 IU

INTERVENTIONS:
Drug: Bemiparin 3500 — Bemiparin sodium 3,500 IU anti Xa/0.2 ml solution for injection in the pre-filled syringe will be provided for each patient in one group; subcutaneously 6 hours after the surgery(orthopedic and non-orthopedic) and then daily for up to 10 days for moderate and high - risk group and for 30 days in very high risk-group patients according to Caprinin risk classification for venous thromboembolism.
  Other Name: Hibor; Laboratories Rovi Pharmaceuticals
  Other Names: Hibor 3500 IU
  Arms: Bemiparin 3500 IU
Drug: Bemiparin 5000 IU — Bemiparin sodium 5000 IU anti Xa/0.2 ml solution for injection in the pre-filled syringe will be provided for each patient in one group; subcutaneously 6 hours after the surgery(orthopedic and non-orthopedic) and then daily for up to 10 days for moderate and high - risk group and for 30 days in very high risk-group patients according to Caprinin risk classification for venous thromboembolism.
  Other Name: Hibor; Laboratories Rovi Pharmaceuticals
  Other Names: Hibor 5000 IU
  Arms: Bemiparin 5000 IU

SUMMARY:
Morbid obesity, is known to be associated with a high risk of VTE and, unfortunately, fixed doses of anticoagulant regimens may not provide optimal VTE prophylaxis in these patients especially after surgery.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is serious and preventable in patients who have undergone recent surgery . Most surgical patients are required to receive VTE prophylaxis, usually pharmacologic prophylaxis. Notwithstanding, rates of appropriate perioperative thromboprophylaxis remain tenaciously low, although the expansion of quality-improvement efforts has led to widespread hospital implementation of prophylaxis strategies.

Obesity, including morbid obesity, is known to be associated with a high risk of VTE and, unfortunately, fixed doses of anticoagulant regimens (unfractionated heparins, low-molecular-weight heparins, and factor Xa inhibitors) may not provide optimal VTE prophylaxis in these patients especially after surgery. Cumulative evidence and works of the literature suggest that anticoagulant dose adjustments in morbidly obese patients may reduce VTE risk. With the increasing rate of morbid obesity, more high-quality clinical trials are needed to prevent VTE in morbidly obese surgical patients providing effective, safe, prevention strategies.

Rationale for Change: Due to challenges in recruiting orthopedic surgical patients within the study timeframe, the protocol has been amended to exclude this patient population. This change ensures the study can proceed with a feasible sample size while maintaining the integrity of the research question regarding LMWH thromboprophylaxis in non-orthopedic surgical patients with morbid obesity. This amendment will not alter the primary research question regarding the efficacy and safety of two doses of LMWH thromboprophylaxis. However, it will narrow the scope of the study to focus exclusively on non-orthopedic surgical patients

ELIGIBILITY:
Inclusion Criteria:

1. Participants required surgical intervention in: general surgery, gynecology, bariatric surgery
2. Moderate, high, and very high risk for venous thromboembolism according to Caprin RAM
3. Participant is willing and able to give informed consent for participation in the study.
4. BMI ≥40kg/m2

Exclusion Criteria:

1. Having any contraindication to LMWH, such as active bleeding, history of heparin-induced thrombocytopenia , baseline platelet count <75 × 108/μl, severe renal disease (glomerular filtration rate <30 ml/minute), severe liver disease, or uncontrolled hypertension (>200/120 mmHg)
2. Known hypersensitivity to unfractionated or LMWHs
3. On oral or parenteral anticoagulants within 5 days before surgery
4. Severe arterial hypertension
5. Unable to comply with the study treatment and/or follow-up
6. Receiving prohibited medications
7. Pregnancy or lactation mother

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with VTE events (Deep vein thrombosis or pulmonary embolism) | up to 30 days after surgery
  Deep vein thrombosis or pulmonary embolism will be confirmed by objective methods (Compression duplex ultrasound for deep vein thrombosis; perfusion/ventilation lung for pulmonary embolism )

SECONDARY OUTCOMES:
Side effects of both Bemiparin doses | up to 30 days after surgery
  Major bleedings,minor bleedings ,total bleeding events (major + minor),thrombocytopenia,injection site reactions, serious adverse events,discontinuations due to adverse side effects

CONTACTS AND LOCATIONS:
Overall Officials: SHAHLA ALALAF, Principal Investigator — Hawler Medical University; Ariana Jawad, Study Chair — Kurdistan Higher Counsel of Medical Specialties; Abdulkader Alany, Study Director — Hawler Medial University; Ali Al-Dabbagh, Study Chair — Hawler Medical University
Locations (1):
- Hawler Medical university, Erbil, Kurdistan Region, Iraq